CLINICAL TRIAL: NCT02986464
Title: Virtual Reality Distraction for Procedural Pain Management in Children With Burn Injuries: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, RN, PhD, Professor, Université de Montréal, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1382
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Burns; Child; Pain
Keywords: Virtual reality; Immersive distraction; Virtual world; Virtual environment; Procedural pain; Acute pain; Pain Management; Children, Child; Kid, Kids; Pediatric, Pediatrics; Young children; Burns; Burn injuries; Burn unit; Hydrotherapy; Burn dressing; Non-pharmacological; Clinical Research; Nursing Practice
MeSH Terms: conditions — Burns; Pain; Pain, Procedural; Acute Pain; Agnosia; Deafness, Autosomal Recessive 1A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pharmacological treatment (Active Comparator)
  Interventions: Other: Standard Pharmacological Treatment
- Virtual Reality distraction (Experimental)
  Interventions: Device: Virtual Reality Prototype

INTERVENTIONS:
Device: Virtual Reality Prototype — VR prototype installed around the tank in the hydrotherapy room to give the child a sense of immersion in the virtual world with a possibility of interaction depending on the child's age and condition.
  Arms: Virtual Reality distraction
Other: Standard Pharmacological Treatment — According to the unit's protocol and adjusted to each participant's age, weight and condition by the anesthetist and the pain clinic nurse.
  Arms: Standard pharmacological treatment

SUMMARY:
Procedural pain is the most intense and often undertreated pain associated with burn injuries. The use of analgesics does not always provide optimal relief and is accompanied by several side effects. Indeed, children with burn injuries still experience severe pain intensity during procedures despite the fact that doses of analgesics used with this population has almost doubled in the last twenty years. Current guidelines on pediatric procedural pain management recommend the combination of non-pharmacological and pharmacological interventions to enhance pain management and decrease the numerous side effects of analgesics. Distraction has been identified among the most effective non-pharmacological interventions for pain as it diverts the child's attention to an attractive element, hindering the perception of the painful stimuli. Virtual reality is a method of active distraction that offers the child a multi-sensory immersive interaction that found many applications for pain management in adult patients. However, very few studies have tested the efficacy of distraction by virtual reality on procedural pain and anxiety in children with burn injuries.

This RCT follows a pilot study (NCT02794103) aimed at assessing the feasibility of a virtual reality prototype developed specifically for the hydrotherapy room of children under seven years old for the relief of procedural pain in children with burn injuries. The aim of the RCT will be to evaluate the effectiveness of the virtual reality prototype in relieving procedural pain in children from 6 months to 7 years old undergoing hydrotherapy session for burn injuries.

DETAILED DESCRIPTION:
BACKGROUND:

Preliminary data from the pilot study showed that the virtual reality prototype installed around the tank in the hydrotherapy room is a feasible and acceptable method of distraction that doesn't interfere with the work of healthcare professionals and could be used as a non-pharmacological method for pain management. A clinical trial is needed to assess the effectiveness of this intervention for procedural pain relief. The pilot study was also informative about the feasibility of the study design and the measurement used. The methods section was modified and adapted consequently for the upcoming trial.

METHODS:

Design: Within-subject/crossover study design. Each child will serve as their own control and will receive both standard and experimental treatment during the same hydrotherapy session through a randomized order.

Sample and Setting: Convenience sampling on the surgical-trauma burn unit at CHU Ste-Justine, of children admitted to the unit or to the day hospital for a burn injury. The intervention will take place in the hydrotherapy room of the CHU Ste-Justine.

Interventions. A) Standard pharmacological treatment as per the unit's protocol. B) VR distraction through the use of a virtual reality prototype installed around the tank in the hydrotherapy room. The prototype has been developed in collaboration with the Society of Arts and Technology (SAT) in Montreal to provide an immersive interactive experience for the burn child in the hydrotherapy tank. The prototype was developed after several meetings between the researchers, the designers and engineers and the surgical trauma team of CHU Ste-Justine. Meetings were followed by an ergonomic study of the hydrotherapy room to meet the unit's and patients' specifications and ensure that it doesn't interfere with the healthcare professionals work.The video games were developed by our team with a personalized care content tailored to the children's developmental stage and to maximize the feeling of immersion and minimize cybersickness, and approved by a team of healthcare professionals in pediatric burn care.

Study proceedings: Hydrotherapy sessions typically last between 20 to 40 minutes. The duration will be divided into two sequences of the same duration (10 to 20 minutes) where the participant receives the same care by the same healthcare professional. For one sequence, only the standard treatment will be administered and for the other sequence, patients will receive the standard treatment in addition to Virtual Reality via the screen around the tank in a randomized order.

Measures: Pain and anxiety measures will be taken before the treatment session at Baseline (T1), in the middle of the first sequence of the session (T2) and in the middle of the second sequence of the session (T3) followed by a measure of healthcare professionals' satisfaction level via a questionnaire developed and pretested by the team after the session (T4). Data will be collected on the average doses of analgesics administered before and during the session, and the side effects experienced.

Data analysis: Quantitative analysis. Mean differences in pain scores between sequences will be compared using Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

* suffer from a burn injury requiring a hydrotherapy session
* presence of a consenting parent who can understand, read and write either French or English

Exclusion Criteria:

* Requiring intensive care
* Having a diagnosed cognitive impairment
* Are unconscious or intubated during the hydrotherapy sessions
* Suffering from epilepsy (considering the nature of the intervention)
* Allergic to opioids or other analgesics used for standard pharmacological treatment
* Having burn injuries on the face preventing them from looking at the VR screen

Will be excluded in posteriori from analysis children sedated for more than 50% of the time during one or both study sequences (score of 3 or 4 on the University of Michigan Sedation Scale).

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Mean Pain Score | T2: 5 minutes within the session (in the middle of the first sequence of the session); T3: 10 minutes within the session (in the middle of the second sequence of the session)
  French version of the Face, Legs, Activity, Cry and Consolability (FLACC)

SECONDARY OUTCOMES:
Mean Pain Score - Observational/Behavioral Complementary measure | T1: baseline; T2: 5 minutes within the session (in the middle of the first sequence of the session); T3: 10 minutes within the session (in the middle of the second sequence of the session)
  Visual Analog Scale by proxy
Comfort | T2: 5 minutes within the session (in the middle of the first sequence of the session); T3: 10 minutes within the session (in the middle of the second sequence of the session)
  Behavioural observation scale of comfort level for child burn victims (OCCEB- BECCO)
Sedation | T1: baseline; T2: 5 minutes within the session (in the middle of the first sequence of the session); T3: 10 minutes within the session (in the middle of the second sequence of the session)
  University of Michigan Sedation Scale (UMSS)
Health professionals' satisfaction level | T4: immediately after the procedure before leaving the hydrotherapy room
  Pre-tested tailored questionnaire including tolerance, positive and negative aspects
Analgesic requirement | T2: 5 minutes within the session (in the middle of the first sequence of the session); T3: 10 minutes within the session (in the middle of the second sequence of the session)
  Rescue dose medication administration

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Khadra, RN, PhD (c), Principal Investigator — Université de Montreal; CHU Ste-Justine Research Center; Sylvie Le May, RN, PhD, Study Director — Université de Montreal; CHU Ste-Justine Research Center
Locations (1):
- CHU Ste. Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khadra C, Ballard A, Paquin D, Cotes-Turpin C, Hoffman HG, Perreault I, Fortin JS, Bouchard S, Theroux J, Le May S. Effects of a projector-based hybrid virtual reality on pain in young children with burn injuries during hydrotherapy sessions: A within-subject randomized crossover trial. Burns. 2020 Nov;46(7):1571-1584. doi: 10.1016/j.burns.2020.04.006. Epub 2020 May 7. PMID 32389349